CLINICAL TRIAL: NCT01103206
Title: Evaluation of a Parathyroid Hormone Suppression Test With Cinacalcet. Comparison: 1- With the Results of the Intravenous Calcium Suppression Test in Healthy Controls; 2- Between Healthy Controls and Patients With Primary Hyperparathyroidism.
Brief Title: Evaluation of a Cincalcet Suppression Test
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009/172/HP
Record Dates: First submitted 2010-04-12; First posted 2010-04-14 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Parathyroid Hormone Suppression Test With Cinacalcet
Keywords: Parathyroid hormone; Cinacalcet; Primary hyperparathyroidism; Diagnosis
MeSH Terms: conditions — Hyperparathyroidism, Primary; Disease | interventions — Cinacalcet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control group (Experimental): Parathyroid hormone suppression tests using successively (each test will be separate for a two week period) an intravenous calcium loading or cinacalcet will be performed in a group of 12 healthy volunteers.
  Interventions: Drug: cinacalcet
- Primary hyperparathyroidism dose I (Experimental): Parathyroid hormone suppression test using the first dose of cinacalcet in patients with primary hyperparathyroidism.
  Interventions: Drug: cinacalcet dose 1
- Primary hyperparathyroidism dose II (Experimental): Parathyroid hormone suppression test in primary hyperparathyroidism using cinacalcet (dose 2).
  Interventions: Drug: cinacalcet dose 2

INTERVENTIONS:
Drug: cinacalcet — Intake of a single tablet of cinacalcet
  Arms: Control group
Drug: cinacalcet dose 1 — PTH suppression test in primary hyperparathyroidism using cinacalcet (dose 1).
  Arms: Primary hyperparathyroidism dose I
Drug: cinacalcet dose 2 — Parathyroid hormone suppression test in primary hyperparathyroidism using cinacalcet (dose 2).
  Arms: Primary hyperparathyroidism dose II

SUMMARY:
The aim of the study is to compare the results of a parathyroid hormone (PTH)suppression test using a single oral tablet of cinacalcet in two groups of subjects: 1- a group of healthy adults in whom the results of the test with cinacalcet will be compared with those of the standardized PTH suppression test with intravenous calcium loading; 2- a group of patients with proven primary hyperparathyroidism in whom the results of the test with cinacalcet will be compared with those obtained during the same test, in healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Control group: healthy adult (>18 years), having signed informed consent, taking no treatment, with effective contraception in unmenopausal women, with normal clinical examination, with normal plasma PTH, calcium, phosphorus, 25 OH vitamin D levels, with normal renal function, with normal 24 hour calciuria.
* Primary hyperparathyroidism group: adult patients (>18 years), having signed informed consent, with effective contraception in unmenopausal women, taking no treatment known to modify calcium-phosphorus status, with normal BMI, in which the diagnosis of primary hyperparathyroidism was confirmed on plasma PTH, calcium, phosphorus, 25 OH vitamin D levels, with normal renal function, with 24 hour calciuria higher than normal.

Exclusion Criteria:

* Control group: significant medical or surgical history, creatinine clearance <60 ml/min, liver insufficiency, arterial hypertension, psychiatric disorder able to modify the compliance to the study, tobacco intoxication, taking a treatment known to modify calcium-phosphorus status, severe known allergy, pregnant women, unmenopaused women without contraception.
* Primary hyperparathyroidism group:secondary hyperparathyroidism, creatinine clearance <60 ml/min, liver insufficiency, psychiatric disorder able to modify the compliance to the study, tobacco intoxication, taking a treatment known to modify calcium-phosphorus status, severe known allergy, pregnant women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Parathyroid hormone suppression test with cainacalcet | Repeated PTH measurements for a period of 12 hours
  Comparison of the plasma parathyroid hormone levels measured in healthy controls during two tests: a test using a single oral dose of cinacalcet and a test using a standardized intravenous calcium loading.

SECONDARY OUTCOMES:
Parathyroid hormone suppression test with cinacalcet in primary hyperparathyroidism | Repeated plasma Parathyroid hormone levels for a period of 12 hours
  Comparison of the results obtained in patients with primary hyperparathyroidism during a cinacalcet suppression test with those obtained using the same test in healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marc J Kuhn, MD, Study Director — University Hospital of Rouen, France:; Anne F Cailleux, MD, Principal Investigator — University Hospital of Rouen, France:
Locations (1):
- University hospital, Rouen, Haute Normandie, France